CLINICAL TRIAL: NCT03962023
Title: Prognostic Impact of Non-invasive Imaging Parameters (Cardiac Echocardiography and MRI) in Patients With Primary Mitral Insufficiency (MI) by Prolapse: Observational Cohort, Monocentric (COHORTE-IM)
Brief Title: Prognostic Impact of Imaging Parameters in Patients With Primary Mitral Insufficiency by Prolapse (COHORTE-IM)
Acronym: COHORTE-IM
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0082
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Mitral Valve Insufficiency
Keywords: Mitral Valve Insufficiency; Imagery; Prognosis
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: Routine follow-up of patients in the Cardiological Functional Explorations department - Valve Disease Centre for their primary mitral insufficiency by prolapse
  Interventions: Other: Echocardiography and MRI

INTERVENTIONS:
Other: Echocardiography and MRI — Analysis of echocardiography and MRI parameters

SUMMARY:
Degenerative mitral insufficiency secondary to valve prolapse is the most common valve disease in Western countries. In the absence of specific treatment, it spontaneously progresses to heart failure and death when it is severe. Surgical mitral valve repair (or mitral plastic surgery) is the preferred treatment for primary mitral insufficiency by prolapse in case of severe leakage if associated with clinical and/or echocardiographic markers of poor prognosis (i.e., with high risk of morbi-mortality during their follow-up).

It is therefore essential to refine the risk stratification of these patients in order to identify at-risk patients who should potentially benefit earlier from invasive care (cardiac surgery), or conversely, close monitoring.

A number of echocardiographic and MRI parameters may have been associated with a poorer prognosis.

A cohort of patients with primary mitral insufficiency (MI) will be followed to study the relationships of a set of factors to patient prognosis.

DETAILED DESCRIPTION:
Degenerative mitral insufficiency secondary to valve prolapse is the most common valve disease in Western countries. In the absence of specific treatment, it spontaneously progresses to heart failure and death when it is severe. Surgical mitral valve repair (or mitral plastic surgery) is the preferred treatment for primary mitral insufficiency by prolapse in case of severe leakage if associated with clinical and/or echocardiographic markers of poor prognosis (i.e., at high risk of morbi-mortality during their follow-up).

It is therefore essential to refine the risk stratification of these patients in order to identify at-risk patients who should potentially benefit earlier from invasive care (cardiac surgery), or conversely, close monitoring.

Beyond the regurgitation severity parameters, a number of regurgitation resonance parameters may have been associated with a poorer prognosis. These parameters include dilation of the left ventricle (increase of telesystolic diameter), of the left atrium, decrease of left ventricular ejection fraction (FE VG), and increase of pulmonary pressures (pulmonary hypertension). The relationship between left, right ventricular function, atrial function evaluated by new echocardiographic techniques (Speckle tracking, 3D) and prognosis has been poorly studied.

These new innovative techniques are now available in clinical routine and allow an evaluation of size and cardiac function parameters in a more reproducible way than conventional methods. The relationship between prognosis and the assessment of regurgitation severity by the convergence zone method (PISA method) has been well documented in the literature. However, the PISA method presents well-documented reproducibility problems. Other methods of quantification exist, either by echocardiography (qualitative, semi-quantitative and quantitative methods) or by MRI (quantitative methods). They are useful in clinical practice in a multiparametric approach, but their relationship to prognosis has been not well studied.

Thus, the prognostic impact of the following parameters must be studied:

* Echocardiographic and MRI parameters of primary insufficiency severity and their combination
* Ventricular and atrial functions measured by innovative echocardiographic methods (speckle tracking, 3D, left ventricular ejection performance parameters)
* The remodeling of cardiac cavities related to mitral insufficiency evaluated by echocardiography and MRI, apart from the diameter of the left ventricle and the size of the left atrium that has already been studied.

A cohort of patients with primary mitral insufficiency (MI) will be followed up to study the relationships of all these factors with patient prognosis. Part of this cohort will be retrospective, and part will be prospective.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with primary mitral insufficiency by prolapse (any grade) diagnosed by Trans-Thoracic Echocardiography (TTE)
* From November 2010 to April 2019 (retrospective cohort)
* From May 2019 to May 2024 (prospective cohort)
* No previous surgery of the mitral valve before the first ultrasound
* Adults
* Patient who has been informed and not opposed to the use of his or her medical record data

Exclusion Criteria:

* Secondary MI
* Primary MI without valve prolapse
* Active endocarditis
* Patient's refusal to participate in the study
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary mitral insufficiency by prolapse, who came or will come to the echocardiography laboratory of Saint Philibert Hospital for a Trans-Thoracic Echocardiography (TTE)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Time before the first morbi-mortality event | 10 years
  The impact of different parameters obtained by Doppler echocardiography (two-dimensional or three-dimensional mode) or MRI on the prognosis of time of the first morbi-mortality event arrival will be studied.
  Morbi-mortality is defined as the occurrence of at least one of the following events during follow-up:
  * Death from any cause
  * Cardiovascular death defined as linked to heart failure, myocardial infarction, arrhythmia episode and sudden death
  * Hospitalization for heart failure
  * Occurrence of atrial fibrillation
  * Occurrence of a stroke

CONTACTS AND LOCATIONS:
Overall Officials: Sylvestre Marechaux, Md, PhD, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic Hospitals, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No